CLINICAL TRIAL: NCT02951013
Title: The Perioperative Liberal or Restrictive Transfusion in Pediatric Liver Transplantation: A Prospective Randomized Controlled Trial
Brief Title: Transfusion Strategies for Pediatric Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLT20161023
Record Dates: First submitted 2016-10-25; First posted 2016-11-01 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Pediatric Patients Who Need Liver Transplantation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- restrictive group (Experimental): Patients in this group will have a transfusion when the hemoglobin concentration falls below 6g/dL, with a target hemoglobin range of 7.5-8.0g/dL.
  Interventions: Other: restrictive transfusion
- liberal group (Active Comparator): Patients in this group will have a transfusion when the hemoglobin concentration falls below 8g/dL, with a target hemoglobin range of 9.5-10.0g/dL.
  Interventions: Other: liberal transfusion

INTERVENTIONS:
Other: restrictive transfusion — Transfusion will start when the hemoglobin concentration falls below 6.0 g/dL
  Arms: restrictive group
Other: liberal transfusion
  Other Names: Transfusion will start when the hemoglobin concentration falls below 8.0 g/dL
  Arms: liberal group

SUMMARY:
The patients assigned to the restrictive group will receive transfusion once the hemoglobin concentration falls below 6.0 g per deciliter, with a target hemoglobin range of 7.5 to 8.0 g per deciliter. Patients assigned to the liberal group will receive transfusion once the hemoglobin concentration falls below 8.0 g per deciliter, with a target hemoglobin range of 9.0 to 10.0 g per deciliter.

The primary outcome: Survival rate in six months after randomization.

Secondary outcomes: Incidence of perioperative complications, including sepsis , pulmonary complications, portal vein thrombosis, hepatic artery thrombosis and transfusion-related adverse events. Intraoperative blood loss, intraoperative blood transfusion amount, postoperative blood transfusion amount in 7 days after surgery, postoperative inflammatory reaction, mechanical ventilation time in the intensive care unit, lengths of stay in the intensive care unit and the hospital，and hospitalization expenses.

ELIGIBILITY:
Inclusion Criteria:

* The investigators study included pediatric patients (the moon's age <36 months) who will receive standard living-donor liver transplantation (LDLT) in Renji Hospital.

Exclusion Criteria:

* The exclusion criteria of the study were a congenital sufferer from heart, lung, kidney, nervous system or blood disease,active Lung infection, a history of liver transplantation, Multivisceral transplantation, refused to participate the study.

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 488 (Estimated)
Dates: Start 2016-12-07 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Survival rate | up to 6 months after randomization

SECONDARY OUTCOMES:
Amount of intraoperative blood transfusion | during surgery
Amount of blood transfusion during perioperative period | up to 7 days after surgery
Heart rate during surgery | during surgery
Blood pressure during surgery | during surgery
Arterial partial pressure of oxygen during surgery | during surgery
Plasma lactic acid concentration during surgery | during surgery
Oxygen uptake rate during surgery | during surgery
Daily score on Pediatric end-stage liver disease (PELD) assessment | up to 7 days after randomization
Length of Mechanical Ventilation in the intensive care unit | at discharge, an average of 2 weeks
Lengths of stay in the intensive care unit | at discharge, an average of 2 weeks
Proportion of patients who need a second hepatic surgery | up to 7 days after randomization
Hospitalization Days | at discharge, an average of 2 weeks
Out of pocket expenditure for hospitalization | at discharge, an average of 2 weeks
Incidence of severe postoperative complications before discharge | from end of surgery till at discharge, an average of 2 weeks
  Postoperative complications include sepsis , pulmonary complications, portal vein thrombosis, hepatic artery thrombosis and transfusion-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Tian, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital affliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided